CLINICAL TRIAL: NCT07349758
Title: DD-PrEP: Pharmacokinetic Evaluation of Single Dosing With Two F/TAF Tablets Among Healthy Volunteers
Brief Title: Evaluation of Single Dosing With Two F/TAF Tablets Among Healthy Volunteers
Acronym: DD-PrEP:
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IRB00488588; DP1DA060602 (NIH)
Record Dates: First submitted 2026-01-15; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Healthy Volunteer; HIV Prevention
Keywords: HIV PrEP; healthy volunteer
MeSH Terms: interventions — tenofovir alafenamide; Emtricitabine; Racivir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- F/TAF dosing (Experimental): Received one-time dosing of two F/TAF tablets
  Interventions: Drug: tenofovir alafenamide [TAF] 50 mg/emtricitabine [FTC] 400mg

INTERVENTIONS:
Drug: tenofovir alafenamide [TAF] 50 mg/emtricitabine [FTC] 400mg — One-time dose of two F/TAF tablets

SUMMARY:
The goal of this study is to evaluate the pharmacokinetics of a one-time dosing of two F/TAF tablets over a 14-day period.

DETAILED DESCRIPTION:
HIV prevention using oral pre-exposure prophylaxis (PrEP) with tenofovir-containing regimens is a promising strategy to reduce the incidence of HIV infection. The study participants will receive a double dose [2 tablets] of Descovy (tenofovir alafenamide [TAF] 25 mg/emtricitabine [FTC] 200mg; F/TAF) and be followed over the course of 14 days. Intensive pharmacokinetic (PK) will occur right after dose administration, and become sparser over the next 14 days. Understanding the PK of TAF, tenofovir (TFV), and FTC and the intracellular metabolites could be used to assess the protective and therapeutic plausibility of alternate, less frequent dosing regimens for PrEP.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age, inclusive on the date of screening
* Provides written informed consent for the study
* Good general health, as determined by medical history, physical examination, vital signs, screening laboratory tests
* Non-reactive HIV test results within four weeks of enrollment
* An estimated glomerular filtration rate (eGFR) of ≥ 70 mL/min/1.73 m2 via the CKD-EPI 2021 eGFRCr equation
* Agrees to use condoms for all sexual events during study participation
* Willing to abstain from oral PrEP use outside of study products for the duration of the study

Exclusion Criteria:

* History of oral PrEP (F/TDF or F/TAF) use in the preceding two months
* Persons who have a reactive or positive HIV result from screening visit.
* Positive hepatitis B surface antigen (HBsAg) test
* Participants with a history of having a gastrectomy, colostomy, ileostomy, or any other procedure altering the gastrointestinal tract or drug absorption
* History of any behaviors that place the participant at high-risk for HIV acquisition (e.g., needle sharing, unprotected sex with ≥1 partner in the prior 2 weeks)
* Taking concomitant medications that that are known inducers/inhibitors of P-gp that would effect TAF absorption
* Pregnancy or lactation
* Any other condition or prior therapy that, in the opinion of the investigator, would preclude informed consent, make study participation unsafe, make the individual unsuitable for the study or unable to comply with the study requirements. Such conditions may include, but are not limited to, current or recent history of severe, progressive, or uncontrolled substance abuse, or renal, hepatic, hematological, gastrointestinal, endocrine, pulmonary, neurological, or cerebral disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Intracellular tenofovir-diphosphate concentrations (fmol/10^6) | 168 hours

CONTACTS AND LOCATIONS:
Overall Officials: Sunil Solomon, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University School of Medicine, Baltimore, Maryland, United States